CLINICAL TRIAL: NCT02718235
Title: Prospective, Multicenter Study to Evaluate the HCCIS as Prognosticator for Overall and Disease-free Survival of Patients After Resection of HCC
Brief Title: Prospective, Multicenter HCCIS Evaluation Study
Acronym: HCCIS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Regensburg (Other)
Collaborators: Else Kröner Fresenius Foundation (Other)
Responsible Party: Principal Investigator, Stefan Brunner, PD Dr. med. Stefan M. Brunner, University of Regensburg
Other Study IDs: HCCIS16
Record Dates: First submitted 2016-03-05; First posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tumor tissue for immunohistochemical analysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Overall survival HCCIS low risk: HCCIS 2 points
  Interventions: Other: Overall survival
- Overall survival HCCIS medium risk: HCCIS 1 point
  Interventions: Other: Overall survival
- Overall survival HCCIS high risk: HCCIS 0 point
  Interventions: Other: Overall survival

INTERVENTIONS:
Other: Overall survival — Observation of overall and disease free survival

SUMMARY:
With this prospective, multicenter trial the investigators aim to establish the Hepatocellular Immune Score (HCCIS), a score that has been developed in a retrospective study, as a new tool for risk stratification of patients after resection of hepatocellular carcinoma that can be widely used in the clinical practice. The investigators expect to show that this score is a prognosticator for overall survival and also disease free survival. Further, it should be demonstrated that the HCCIS is a risk stratification tool that is independent from clinical or descriptive parameters. Additionally, the investigators plan to elucidate that the respective HCCIS risk groups are not only different with respect to immunological infiltration but are also different with respect to tumor biology. The finding, that tumors of the respective risk groups show different tumor biology leads to the assumption that different therapy strategies need to be applied. Therefore, in a translational approach we aim to build up a data base with HCC tumor organoids and test the effect of CD8+IL-33+ effector-memory cells on HCC tumor organoids of the respective HCCIS risk groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old who are receiving primary liver resection in curative intent for HCC after informed consent is obtained.

Exclusion Criteria:

* Patients who have not given informed consent or who have withdrawn their consent will be excluded from this analysis. In case there is not enough liver tissue for a histological analysis or the remaining liver tissue is not enough to perform a routine pathological analysis patients have to be excluded from the further analysis. In case of an R1 or R2 resection, patients have to be excluded from further analysis. However, these patients will remain in the study as an intention to treat analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >18 years old who are receiving primary liver resection in curative intent for HCC after informed consent is obtained.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-06; Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
The HCC immune score (HCCIS) is a survival prognosticator of patients after liver resection for HCC | 3 years
  Overall survival

SECONDARY OUTCOMES:
The HCC immune score (HCCIS) to prognosticate disease free survival of patients after liver resection for HCC | 3 years
  Disease free survival

CONTACTS AND LOCATIONS:
Overall Officials: Stefan M Brunner, MD, Principal Investigator — Department of Surgery, University Medical Center Regensburg, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: No